CLINICAL TRIAL: NCT05728957
Title: A Prospective Diagnostic Cohort Study to Compare the Accuracy of Renal Mass Biopsy, PEER, and 99mTc-sestamibi SPECT/CT for Patients With Clinically Localized Renal Tumors
Brief Title: Renal Mass Biopsy, PEER, and 99mTc-sestamibi SPECT/CT for Patients With Clinically Localized Renal Tumors
Acronym: BIOPSy
Status: Recruiting | Type: Observational
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Hiten Patel, Affiliate Assistant Professor, Loyola University
Other Study IDs: 215278
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Kidney Tumor; Renal Benign Neoplasm; Renal Malignant Tumor
Keywords: Kidney Tumor; Survey Questions; Benign; Malignant; Renal Benign Neoplasm; Renal Malignant Tumor; Nuclear Imaging; Computed Tomography
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Urine, and/or Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to better tell apart whether kidney tumors are benign (not cancer) or malignant (cancer) based on a biopsy or imaging tests and ask patients how they feel about decisions they make about treatment of their kidney tumor.

The main objectives are:

To estimate and compare the diagnostic accuracy of renal mass biopsy alone, PEER (with renal mass biopsy), and 99mTc-sestamibi SPECT/CT (with renal mass biopsy for hot tumors) to differentiate malignant and benign renal tumors.

To estimate and compare the diagnostic accuracy of renal mass biopsy, PEER (with renal mass biopsy), and 99mTc-sestamibi SPECT/CT (with renal mass biopsy for hot tumors) to differentiate oncocytoma from chromophobe RCC.

Participants will be asked to complete survey questions related to their health and kidney tumor at the start and end of the study. These can be done on paper, electronically, or by telephone.

DETAILED DESCRIPTION:
The investigators are asking the participant to take part in this research study because they were diagnosed with a kidney tumor. Kidney tumors can be benign (not cancer) or malignant (cancer) and the investigators hope to figure out how to better tell them apart before surgery or other treatment.

The investigators hope to better tell apart whether kidney tumors are benign (not cancer) or malignant (cancer) based on a biopsy or imaging tests and ask patients how they feel about decisions they make about treatment of their kidney tumor.

Biopsy is a standard test to determine if a tumor is cancerous before making a treatment decision.

The imaging test (99mTc-sestamibi SPECT/CT) the investigators are studying has been studied before and found to help identify benign kidney tumors. It is not approved by the Food and Drug Administration (FDA) for imaging kidney tumors. It is FDA approved for use in imaging the heart and breasts. It has been studied for use in parathyroid gland imaging.

The participant will be asked to complete survey questions related to their health and kidney tumor at the start and end of the study. The participant will receive a 99mTc-sestamibi SPECT/CT scan (if they have not had one already) for research purposes. The participant will receive a biopsy of the kidney tumor (if they have not had one already) as part of their routine clinical care. The participant will then receive treatment of the kidney tumor as determined by consultation with their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with a clinically localized (cT1) renal tumor ≤7cm in size with a solid component suspicious for malignancy based on cross-sectional imaging
* Pre-existing CT images of the mass with and without contrast or planned CT to ensure both with and without contrast images of the mass have been obtained within a 365-day window
* Participants must be greater than or equal to 18 years of age
* Eligible or planned to undergo partial or radical nephrectomy as determined by primary urologist
* Eligible or planned to receive renal mass biopsy as determined by primary urologist
* Estimated glomerular filtration rate of ≥30 ml/min/1.73 m2 as calculated by the CKD-EPI (Chronic Kidney Disease-Epidemiology Collaboration) Equation

Exclusion Criteria:

* Participants must not be pregnant (as determined by local policy by radiology / imaging center)
* Participants must not have evidence of clinical nodal or distant metastasis.
* Participants must not have had a history of other malignancy with concern for renal metastasis.
* Participants must not have any known allergy to technetium or sestamibi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be 18 years of age and older, male or female and diagnosed with a kidney tumor. Kidney tumors can be benign (not cancer) or malignant (cancer).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-02 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Histologic Classification (malignant vs. benign) | Until surgical extirpation or 1 year repeat biopsy
  The classification of each tumor as malignant or benign by the diagnostic approaches of interest will be compared to the primary endpoint of malignant vs. benign based on surgical pathology or biopsy.

SECONDARY OUTCOMES:
Histologic Classification (RCC vs. oncocytoma) | 30 days after surgical extirpation or 1 year repeat biopsy
  The classification of each tumor as RCC or oncocytoma by the diagnostic approaches of interest will be compared to the primary endpoint of RCC vs. oncocytoma based on surgical pathology or biopsy.
Non-diagnostic rate for renal mass biopsy | 30 days after surgical extirpation or 1 year repeat biopsy
  To estimate the non-diagnostic rate of renal mass biopsy.
Patient-reported measures/outcomes related to mental health, physical health, distress, and regret | 30 days after surgical extirpation or 1 year repeat biopsy
  To describe patient-reported measures/outcomes related to mental health, physical health, distress, and regret for the diagnosis and management of renal tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Hiten D Patel, MD, MPH, Principal Investigator — Loyola University; Gopal N Gupta, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No